CLINICAL TRIAL: NCT00297297
Title: Preoperative Selection of Solitary Solid Cold Thyroid Nodules - A Prospective Study on the Value of Sonography, Cytology, Immunostaining and Molecular Profiling
Brief Title: Improved Preoperative Selection of Cold Thyroid Nodules
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Herlev Hospital (Other)
Responsible Party: Finn N Bennedbaek, Md, PhD (principal investigator), Herlev University Hospital
Other Study IDs: HH-FB-10
Record Dates: First submitted 2006-02-27; First posted 2006-02-28 (Estimated); Last update posted 2010-02-25 (Estimated); Status verified 2007-10

CONDITIONS: Thyroid Nodules
Keywords: Solitary solid and scintigraphically cold thyroid nodules
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Other: No intervention. Applying gene profiling on needle aspirates
  Other Names: Genetics - molecular profiling of tissue samples

SUMMARY:
Molecular gene profiling of fine-needle aspiration samples in addition to fine-needle aspiration cytology can improve the selection of patients with benign versus malignant thyroid nodules with improved sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Solitary thyroid nodules that appear solid on ultrasound and cold on a scintiscan

Exclusion Criteria:

* Pregnancy and lactation
* Age below 20 years

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary referral center (Endocrine outpatient - University Hosiptal - clinic). Patients referred with a solitary thyroid nodule
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-12; Study Completion 2011-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Finn N Bennedbaek, MD, PhD, Principal Investigator — Department of Endocrinology and Metabolism, Herlev University Hospital, DK-2730 Herlev, Denmark
Locations (1):
- Outpatient clinic of The Department of Endocrinology, Herlev University Hospital, Copenhagen, Denmark

REFERENCES:
- [Result] Finley DJ, Zhu B, Barden CB, Fahey TJ 3rd. Discrimination of benign and malignant thyroid nodules by molecular profiling. Ann Surg. 2004 Sep;240(3):425-36; discussion 436-7. doi: 10.1097/01.sla.0000137128.64978.bc. PMID 15319714